CLINICAL TRIAL: NCT00174460
Title: Somatropin Therapy For Short Children Born Of Premature Gestation, A Controlled, Prospective Randomized, Multicenter Study With An Untreated Control Group.
Brief Title: Somatropin Therapy In Children Born Preterm But Appropriate For Gestational Age
Acronym: AGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6281273
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-05-12 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Growth Hormone Therapy; Infant, Very Low Birth Weight
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Active Comparator)
  Interventions: Drug: Somatropin; Other: Control Arm
- Control Arm (No Intervention)

INTERVENTIONS:
Drug: Somatropin — Controlled, prospective, randomized, multicenter study with an untreated (control) group during the first year. The children will be randomized into treatment or untreated (control) group. After one year the control group will undergo GH-therapy, too. Children randomized to the control group will get the possibility to continue treatment for a further year. The study will end after 2 and 3 years of observation, respectively.
  Arms: Treatment Arm
Other: Control Arm — Controlled, prospective, randomized, multicenter study with an untreated (control) group during the first year. The children will be randomized into treatment or untreated (control) group. After one year the control group will undergo GH-therapy, too. The study will end after 2 and 3 years of observation, respectively. Children randomized to the control group will get the possibility to continue treatment for a further year.
  Arms: Treatment Arm

SUMMARY:
Safety and efficacy of Somatropin will be evaluated in short children born with a list weight below 1500 g and that did not catch up to normal height at the age of 4.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

* Prepubertal caucasian boys between 4 and 10 years of age and girls between 4 and 9 years of age.
* Girls: Tanner stage 1 breast development
* Boys: Testis volume <= 3ml
* Tanner stage 1 pubic hair development (to exclude confounding effect of adrenarche on growth velocity, insulin sensitivity and body composition).
* (In case of any signs or symptoms of gonadal puberty a GnRH-Test must decide if the subject is still pubertal.)
* Height <=-2 SD for chronological age (Brandt/Reinken).
* Growth velocity SDS below 0 SD for chronological age (Brandt/Reinken based on 12+/- 3 months observation period before screening).
* Premature born defined as <=1500 g birth weight.
* GH sufficiency (GH level > 7 ug/l following any routine GH stimulation test).
* Written informed consent of both parents (legal guardians) and oral/written consent of subject due to age specific information.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

* Other endocrine diseases except for well substituted hypothyroidism.
* Severe chronic diseases or medication that might influence linear growth or insulin sensitivity (e.g. Glucocorticoids).
* Positive GAD and IA-2 antibodies (for type 1 diabetes).
* History of malignancy
* Children who meet all of the following 4 criteria:
* actual body height < -2,5 SDS (Brandt/Reinken) and parent adjusted target height < -1 SDS (Hermanussen and Cole, 2003)
* length and/or body weight retardations adjusted to gestational age at birth < -2,0 SDS (Lawrence et al., 1989, Voigt et al., 1996)
* children with chronological age > = 4 years and
* growth velocity < 0 SDS during the last year before inclusion.
* Chromosomal aberrations or syndromes.
* Suspected non-compliance or impossibility to follow the two or three year treatment schedule, respectively (e.g. social implications).
* Severe hemiparesis and severe CNS defects
* Retinopathia > third degree or laser treatment as newborns.
* Participation in any other clinical trial during active treatment phase.
* Other severe acute or chronic medical or psychiatric condition or clinically relevant laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Germany (8):
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Homburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Tübingen

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281273&StudyName=Somatropin%20Therapy%20In%20Children%20Born%20Preterm%20But%20Appropriate%20For%20Gestational%20Age

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin: The children were randomized into a treated group receiving 0.068 mg/kg/day (0.48mg/kg/week) subcutaneous somatropin according to exact body weight specific calculation. Dose adjustments were made at 6 month intervals. (mg=milligrams, kg=kilograms)
- Control Arm: The children were randomized into control group and after 1 year underwent Growth Hormone (GH) therapy, with 0.068 mg/kg/day (0.48mg/kg/week) subcutaneous somatropin according to exact body weight specific calculation. Dose adjustments were made at 6 month intervals. mg=milligram, kg=kilogram.
Period: Overall Study
Arm/Group | Somatropin | Control Arm
Started | 18 | 15
Received Study Treatment | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Somatropin | Control Arm | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.4 (1.6) | 5.7 (1.9) | 5.5 (1.7)
Age, Customized [Number; unit: Participants] — 1 subject in each treatment group was below the age of 4 at screening. However, both of them were 4 years old when treatment began; they did not violate the corresponding inclusion criterion.
  Participants
    <4 years | 1 (1.5) | 1 (1.9) | 2 (1.7)
    ≥4 years and <8 years | 14 | 11 | 25
    ≥8 years and <12 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Height Standard Deviation Score (SDS) After 1 Year
Description: Change in Height SDS after 1 year where SDS=height minus mean (age-and sex-matched reference) divided by SD (age and sex-matched reference).
Time Frame: Baseline to 1 year (Month 12)
Population: Full Analysis Set (FAS; all randomized subjects who had at least 1 post-baseline efficacy measurement); Control group received Somatropin from Month 12 onwards.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters | 1.099 (0.0714) | 0.108 (0.0783)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from analysis of covariance method (ANCOVA) adjusted for baseline height SDS and target height SDS; Last observation carried forward (LOCF); Mean Difference (Final Values) = 0.991, 95% CI 2-sided [0.773 to 1.210], Standard Error of Mean 0.1067

2. Secondary Outcome: Change From Baseline in Growth Velocity After 1 Year and After 2 Years
Description: Growth velocity measured as centimeters per year.
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards.
Measure: Least Squares Mean (Standard Error); unit: centimeters per year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters per year
  Month 12 | 5.110 (0.2623) | 0.695 (0.2881)
  Month 24 | 3.049 (0.3546) | 3.934 (0.3893)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from ANCOVA adjusted for baseline growth velocity, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = 4.415, 95% CI 2-sided [3.605 to 5.225], Standard Error of Mean 0.3950
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.108, ANCOVA; Results from ANCOVA adjusted for baseline growth velocity, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = -0.884, 95% CI 2-sided [-1.977 to 0.208], Standard Error of Mean 0.5327

3. Secondary Outcome: Change From Baseline in Growth Velocity SDS After 2 Years
Description: Change in Growth Velocity SDS after 2 years (24 months) where SDS = growth velocity minus mean (age-and sex-matched reference) divided by SD (age and sex-matched reference).
Time Frame: Baseline, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards.
Measure: Least Squares Mean (Standard Error); unit: centimeters per year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters per year | 4.751 (0.4716) | 5.825 (0.5177)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference; Test type: Superiority or Other; p = 0.141, ANCOVA; Results from ANCOVA adjusted for baseline growth velocity SDS and target height SDS; LOCF; Mean Difference (Final Values) = -1.074, 95% CI 2-sided [-2.524 to 0.376], Standard Error of Mean 0.7089

4. Secondary Outcome: Change From Baseline in Height After 1 Year and After 2 Years
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters
  Month 12 | 10.467 (0.2439) | 5.927 (0.2677)
  Month 24 | 18.908 (0.6507) | 14.844 (0.7149)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from ANCOVA adjusted for baseline height, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = 4.540, 95% CI 2-sided [3.789 to 5.291], Standard Error of Mean 0.3661
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from ANCOVA adjusted for baseline height, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = 4.064, 95% CI 2-sided [2.049 to 6.080], Standard Error of Mean 0.9822

5. Secondary Outcome: Change From Baseline in Height SDS After 2 Years
Description: Change in Height SDS after 2 years (24 months) where SDS = height minus mean (age-and sex-matched reference) divided by SD (age and sex-matched reference).
Time Frame: Baseline, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters | 1.710 (0.1075) | 0.991 (0.1179)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from ANCOVA adjusted for baseline height SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.719, 95% CI 2-sided [0.390 to 1.047], Standard Error of Mean 0.1606

6. Secondary Outcome: Change From Baseline in Body Composition (Skinfold Thickness) After 1 Year and After 2 Years: Triceps
Description: Body composition measured as skinfold thickness at tricep in millimeters (mm); measured halfway down the left upper arm with arm hanging in relaxed position at participant's side.
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards. N=number of participants with evaluable data at observation.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
millimeters
  Month 12 | -2.20 (0.341) | 0.50 (0.353)
  Month 24 | -1.30 (0.511) | -0.83 (0.548)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from ANCOVA adjusted for baseline skinfold thickness, target height SDS, age, and sex; LOCF; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-3.73 to -1.68], Standard Error of Mean 0.497
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.537, ANCOVA; Results from ANCOVA adjusted for baseline skinfold thickness, target height SDS, age, and sex; LOCF; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-2.04 to 1.09], Standard Error of Mean 0.758

7. Secondary Outcome: Change From Baseline in Body Composition (Skinfold Thickness) After 1 Year and After 2 Years: Subscapular
Description: Body composition measured as subscapular skinfold thickness in millimeters (mm); measured laterally just below the angle of the left scapula.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
millimeters
  Month 12 | 0.08 (0.276) | 0.46 (0.286)
  Month 24 | 0.27 (0.231) | 0.50 (0.247)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.364, ANCOVA; Results from ANCOVA adjusted for baseline skinfold thickness, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.21 to 0.46], Standard Error of Mean 0.405
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.506, ANCOVA; Results from ANCOVA adjusted for baseline skinfold thickness, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.94 to 0.48], Standard Error of Mean 0.345

8. Secondary Outcome: Change From Baseline in Body Composition (Skinfold Thickness) After 1 Year and After 2 Years: Suprailiac
Description: Body composition measured as suprailiac skinfold thickness in millimeters (mm); measured just above the iliac crest in the middle-axillary line.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
millimeters
  Month 12 | 0.51 (0.783) | 0.45 (0.849)
  Month 24 | 0.90 (0.688) | 0.79 (0.774)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.959, ANCOVA; Results from ANCOVA adjusted for baseline skinfold thickness, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-2.42 to 2.54], Standard Error of Mean 1.188
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.919, ANCOVA; Results from ANCOVA adjusted for baseline skinfold thickness, target height SDS, sex, and age; LOCF; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-2.11 to 2.32], Standard Error of Mean 1.065

9. Secondary Outcome: Change From Baseline in Volumetric Cortical Bone Mineral Density (BMD) Using Peripheral Quantitative Computed Tomography (pQCT) After 1 Year and After 2 Years
Description: Volumetric Cortical BMD measured as milligrams per cubic millimeter (mg/mm3). BMD (proximal radius) SDS (number of standard deviations a participant's BMD differs from the average BMD of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards; (n)=number of participants from FAS with evaluable pQCT data for somatropin and control arm groups, respectively.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
z-score
  Month 12 (n=2, 6) | -1.055 (0.6802) | -0.162 (0.3600)
  Month 24 (n=2, 6) | 0.284 (0.5023) | -0.433 (0.2658)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.336, ANCOVA; Results from ANCOVA adjusted for baseline volumetric cortical bone mineral density SDS and target height SDS; LOCF; Mean Difference (Final Values) = -0.892, 95% CI 2-sided [-3.158 to 1.374], Standard Error of Mean 0.8161
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.300, ANCOVA; Results from ANCOVA adjusted for baseline volumetric cortical bone mineral density SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.717, 95% CI 2-sided [-0.956 to 2.391], Standard Error of Mean 0.6027

10. Primary Outcome: Change in Growth Velocity Standard Deviation Score (SDS) After 1 Year
Description: Change in Growth Velocity (GV) SDS after 1 year where SDS=GV minus mean (age-and sex-matched reference) divided by SD (age and sex-matched reference).
Time Frame: Baseline to 1 year (Month 12)
Population: FAS; Control group received Somatropin from Month 12 onwards.
Measure: Least Squares Mean (Standard Error); unit: centimeters per year
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters per year | 7.117 (0.4384) | 1.502 (0.4814)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference; Test type: Superiority or Other; p < 0.001, ANCOVA; Results from ANCOVA adjusted for baseline growth velocity SDS and target height SDS; LOCF; Mean Difference (Final Values) = 5.615, 95% CI 2-sided [4.266 to 6.963], Standard Error of Mean 0.6591

11. Secondary Outcome: Change From Baseline in Bone Structure Using pQCT After 1 Year and 2 Years: Cortical Cross-sectional Area (CSA)
Description: Bone structure Cortical CSA measured as millimeters squared (mm2). CSA (proximal radius) SDS (number of standard deviations a participant's CSA differs from the average CSA of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
z-score
  Month 12 (n=2, 5) | -0.465 (0.7799) | 0.017 (0.4559)
  Month 24 (n=2, 6) | -0.595 (0.7462) | 0.609 (0.3907)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.653, ANCOVA; Results from ANCOVA adjusted for baseline cortical cross-sectional area SDS and target height SDS; LOCF; Mean Difference (Final Values) = -0.482, 95% CI 2-sided [-3.558 to 2.595], Standard Error of Mean 0.9666
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.251, ANCOVA; Results from ANCOVA adjusted for baseline cortical cross-sectional area SDS and target height SDS; LOCF; Mean Difference (Final Values) = -1.205, 95% CI 2-sided [-3.701 to 1.292], Standard Error of Mean 0.8991

12. Secondary Outcome: Change From Baseline in Bone Structure Using Peripheral Quantitative Computed Tomography (pQCT) After 1 Year and 2 Years: Total Cross-sectional Area (CSA)
Description: Bone structure Total CSA measured as millimeters squared (mm2). Total CSA (proximal radius) SDS (number of standard deviations a participant's CSA differs from the average CSA of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
z-score
  Month 12 (n=2, 5) | 0.375 (0.9345) | 0.239 (0.5537)
  Month 24 (n=2, 6) | 0.243 (0.3694) | -0.049 (0.1955)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.914, ANCOVA; Results from ANCOVA adjusted for baseline total cross-sectional area SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.135, 95% CI 2-sided [-3.524 to 3.795], Standard Error of Mean 1.1499
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.547, ANCOVA; Results from ANCOVA adjusted for baseline total cross-sectional area SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.292, 95% CI 2-sided [-0.939 to 1.522], Standard Error of Mean 0.4432

13. Secondary Outcome: Change From Baseline in Bone Structure Using pQCT After 1 Year and 2 Years: Muscle Cross-sectional Area (CSA)
Description: Bone structure Muscle CSA measured as millimeters squared (mm2). CSA (proximal radius) SDS (number of standard deviations a participant's CSA differs from the average CSA of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
z-score
  Month 12 (n=2, 6) | 2.084 (0.3628) | -0.227 (0.1688)
  Month 24 (n=2, 6) | 2.402 (0.5221) | 0.776 (0.2428)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.007, ANCOVA; Results from ANCOVA adjusted for baseline muscle cross-sectional area SDS and target height SDS; LOCF; Mean Difference (Final Values) = 2.310, 95% CI 2-sided [1.049 to 3.572], Standard Error of Mean 0.4542
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.068, ANCOVA; Results from ANCOVA adjusted for baseline muscle cross-sectional area SDS and target height SDS; LOCF; Mean Difference (Final Values) = 1.626, 95% CI 2-sided [-0.189 to 3.440], Standard Error of Mean 0.6536

14. Secondary Outcome: Change From Baseline in Bone Structure Using pQCT After 1 Year and 2 Years: Cortical Thickness (CT)
Description: Cortical Thickness measured as millimeters (mm). CT (proximal radius) SDS (number of standard deviations a participant's CT differs from the average CT of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards. Cortical thickness was not analyzed as planned.
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in Bone Structure Using pQCT After 1 Year and 2 Years: Marrow Area (MA)
Description: Marrow Area measured as millimeters squared (mm2). MA (proximal radius) SDS (number of standard deviations a participant's MA differs from the average MA of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards. Marrow Area was not analyzed as planned.
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Bone Stability Using pQCT After 1 Year and After 2 Years: Strength-strain Index (SSI)
Description: Bone stability expressed as polar SSI in cubic millimeters (mm3). SSI (proximal radius) SDS (number of standard deviations a participant's SSI differs from the average SSI of their age and sex). Baseline and post-baseline SDS values transformed to age and sex specific z-score (Ln(test result/M)]/S); Ln=natural logarithm; M=age- or height-) and sex-specific mean value; S=age-(or height-) and sex-specific coefficient of variation) then change from baseline is calculated. Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
z-score
  Month 12 (n=2, 6) | 0.648 (0.4224) | 0.088 (0.2243)
  Month 24 (n=2, 6) | 0.477 (0.3925) | 0.363 (0.2084)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.331, ANCOVA; Results from ANCOVA adjusted for baseline strength-strain index SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.560, 95% CI 2-sided [-0.846 to 1.965], Standard Error of Mean 0.5061
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.820, ANCOVA; Results from ANCOVA adjusted for baseline strength-strain index SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [-1.192 to 1.420], Standard Error of Mean 0.4703

17. Secondary Outcome: Change From Baseline in Muscle Strength: Hand Grip SDS After 1 Year and After 2 Years
Description: Muscle strength determined by measuring grip force (kilograms) using hand grip dynamometer for participants ≥6 years of age. Baseline and post-baseline SDS values transformed to age and sex specific z-score. Change in hand grip calculated as SDS where SDS = hand grip minus mean (age- and sex-matched reference) divided by SD (age- and sex-matched reference). Positive values are above the average for participant's age and sex; negative values are below the average.
Time Frame: Baseline, Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards; (n)=number of participants ≥6 years of age with evaluable data at observation for Somatropin and Control Arm, respectively. SDS reference values used were for the right hand but the hand grip strength measured for this study was for the dominant hand (may not have been the right hand).
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
z-score
  Month 12 (n=7, 5) | 0.37 (0.268) | 0.28 (0.318)
  Month 24 (n=7, 6) | 1.14 (0.218) | 0.92 (0.236)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p = 0.844, ANCOVA; Results from ANCOVA adjusted for baseline hand grip strength SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.88 to 1.05], Standard Error of Mean 0.420
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p = 0.519, ANCOVA; Results from ANCOVA adjusted for baseline hand grip strength SDS and target height SDS; LOCF; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.52 to 0.96], Standard Error of Mean 0.329

18. Secondary Outcome: Number of Participants With Change in Insulin Sensitivity: Somatropin
Description: Insulin sensitivity calculated as incidence of pathological glucose intolerance assessed prior to randomization (Screening Day -3 to Baseline Day 0) and at final visit (final visit: Somatropin treatment group=Month 24). Pathological glucose intolerance (oral glucose tolerance test) measured as venous (blood or plasma) with range minimum 120 milligrams per deciliter (mg/dL) to >140 mg/dL; capillary (blood) with range minimum 120 mg/dL to >120 mg/dL; or method not known with range minimum 120 mg/dL to >120 mg/dL.
Time Frame: Baseline, Month 24
Population: FAS
Measure: Number; unit: participants
Arm/Group | Somatropin
Number analyzed (Participants) | 18
participants
  Baseline: tolerant | 18
  Baseline: intolerant | 0
  Month 24: tolerant | 16
  Month 24: intolerant | 0

19. Secondary Outcome: Number of Participants With Change in Insulin Sensitivity: Control Arm
Description: Insulin sensitivity calculated as incidence of pathological glucose intolerance assessed prior to randomization (Screening Day -3 to Baseline Day 0) and at final visit (final visit: Control Arm=Month 36). Pathological glucose intolerance (oral glucose tolerance test) measured as venous (blood or plasma) with range minimum 120 milligrams per deciliter (mg/dL) to >140 mg/dL; capillary (blood) with range minimum 120 mg/dL to >120 mg/dL; or method not known with range minimum 120 mg/dL to >120 mg/dL.
Time Frame: Baseline, Month 36
Population: FAS; Control group received Somatropin from Month 12 onwards.
Measure: Number; unit: participants
Arm/Group | Control Arm
Number analyzed (Participants) | 15
participants
  Baseline: tolerant | 14
  Baseline: intolerant | 1
  Month 36: tolerant | 11
  Month 36: intolerant | 2

20. Secondary Outcome: Growth Curve Comparison Based on Height SDS
Description: Growth curve comparison with height SDS in centimeters as the dependent variable; SDS = height minus mean (age-and sex-matched reference) divided by SD (age and sex-matched reference).
Time Frame: Month 12, Month 24
Population: FAS; Control group received Somatropin from Month 12 onwards. Data for Month 36 (applicable only to the Control Arm) is reported in a separate outcome measure.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters
  Month 12 | -2.260 (0.0735) | -3.259 (0.0802)
  Month 24 | -1.638 (0.1016) | -2.327 (0.1122)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p < 0.001, Mixed models analysis; Results from repeated measures mixed models analysis adjusted for baseline height SDS, visit, visit*treatment and target height SDS; Mean Difference (Final Values) = 0.998, 95% CI 2-sided [0.778 to 1.219], Standard Error of Mean 0.1095
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p < 0.001, Mixed models analysis; [statistical method as in outcome 20, analysis 1]; Mean Difference (Final Values) = 0.688, 95% CI 2-sided [0.382 to 0.994], Standard Error of Mean 0.1519

21. Secondary Outcome: Growth Curve Comparison Based on Height SDS: Control Arm
Description: Growth curve comparison with height SDS in centimeters as the dependent variable; SDS = height minus mean (age-and sex-matched reference) divided by SD (age and sex-matched reference). Control Arm final visit=Month 36.
Time Frame: Month 36
Population: FAS; Control group received Somatropin from Month 12 onwards. N=number of subjects with evaluable data at observation. Month 36 visit not applicable to Somatropin treatment group.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Control Arm
Number analyzed (Participants) | 14
centimeters | -1.794 (0.1318)

22. Secondary Outcome: Growth Curve Comparison Based on Height
Description: Growth curve comparison with height in centimeters as the dependent variable.
Time Frame: Month 12, Month 24
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Somatropin | Control Arm
Number analyzed (Participants) | 18 | 15
centimeters
  Month 12 | 114.228 (0.3330) | 109.644 (0.3733)
  Month 24 | 123.351 (0.4830) | 119.788 (0.5255)
Statistical Analysis 1: Comparison: Somatropin vs Control Arm; Treatment difference Month 12; Test type: Superiority or Other; p < 0.001, Mixed models analysis; Results from repeated measure mixed models analysis adjusted for baseline height, sex, age, visit, visit*treatment and target height SDS; Mean Difference (Final Values) = 4.585, 95% CI 2-sided [3.806 to 5.363], Standard Error of Mean 0.3859
Statistical Analysis 2: Comparison: Somatropin vs Control Arm; Treatment difference Month 24; Test type: Superiority or Other; p < 0.001, Mixed models analysis; [statistical method as in outcome 22, analysis 1]; Mean Difference (Final Values) = 3.563, 95% CI 2-sided [2.134 to 4.992], Standard Error of Mean 0.7080

23. Secondary Outcome: Growth Curve Comparison Based on Height: Control Arm
Description: Growth curve comparison with height in centimeters as the dependent variable.
Time Frame: Month 36
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Control Arm
Number analyzed (Participants) | 14
centimeters | 128.049 (0.7821)

ADVERSE EVENTS:
Description: Safety population=all participants who received at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Somatropin | Control Arm
Serious Adverse Events (participants affected / at risk) | 5/18 | 1/15
Other Adverse Events (participants affected / at risk) | 13/18 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin (N=18) | Control Arm (N=15)
Pyrexia (General disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Facial palsy (Nervous system disorders) | 0 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somatropin (N=18) | Control Arm (N=15)
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Visual impairment (Eye disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 1 | 2
Ear infection (Infections and infestations) | 1 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 2
Scarlet fever (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 4 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Varicella (Infections and infestations) | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis allergic (Musculoskeletal and connective tissue disorders) | 1 | 0
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Attention deficit / hyperactivity disorder (Psychiatric disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Result values for the primary outcome measures were revised at the final analysis due to programmatic corrections: age rounded up if >6 months past last birthday. Height and height SDS not rounded for final analysis; rounded only for the reports.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.